CLINICAL TRIAL: NCT03499379
Title: Effect of Initiation of Intrauterine Contraception on Hair Cortisol Concentration
Brief Title: Stress Hormones and IUDs
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Nora Doty, MD, Instructor, Oregon Health and Science University
Other Study IDs: OHSU IRB 18244
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Contraception; Mood Change
Keywords: Intrauterine device (IUD); Depression; Stress hormones; Mood changes
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A hair sample of approximately 10 (up to 20) hairs cut close to the scalp of the posterior vertex.
  Whole blood samples collected at each study visit (approximately 10mL). The serum from those samples will tested for hormone levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women initiating use of an intrauterine device: Women obtaining a copper or hormonal intrauterine device for the purpose of contraception.
  A hair sample of approximately 10 (up to 20) hairs cut close to the scalp of the posterior vertex will be taken at the time of IUD insertion, 6 months post-insertion, and 12 months post-insertion.
  Interventions: Device: Mirena; Device: Paraguard

INTERVENTIONS:
Device: Mirena — A radio-opaque T-shaped polyethylene device containing 52mg of levonorgestrel dispersed in polydimethylsiloxane on its stem. The progestin is released at a rate of 15 mcg per day.
  Other Names: levonorgestrel intrauterine system
Device: Paraguard — A T-shaped polyethylene device with 380 mm2 of exposed surface area of fine copper wire wound around its arms and stem. Barium sulfate has been added to the polyethylene frame to make the device radio-opaque. A 3-mm plastic ball is located at the base of the IUD, through which the polyethylene monofilament string passes.
  Other Names: Copper T380A IUD

SUMMARY:
Determine what kind of side effects women experience in the first year after they start using an intrauterine device.

DETAILED DESCRIPTION:
The purpose of this study is to find out if there is a difference in levels of stress hormones in women who use copper or hormonal intrauterine devices (IUDs). This study will provide more information on the potential effect of levonorgestrel intrauterine system (LNG-IUS) use on an individual's stress response. Ultimately, this study hopes to provide data to better counsel women on potential mood effects of the LNG-IUS. From a research and clinical management perspective, hair cortisol may provide a tool to evaluate women at risk for discontinuation of hormonal contraception due to concern of mood symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy
* Age 18-39 years
* Regular menstrual cycles
* Getting an IUD for the purpose of contraception

Exclusion Criteria:

* History of mood disorders
* BMI less than 18.5 or greater than 35
* Chronic medical conditions
* Recently pregnant or lactating

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study participants will be selected from women's health care clinics in the community.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Mean change in hair cortisol concentration - 6 months | Baseline & 6 months post-insertion
  A hair sample of approximately 10 (up to 20) hairs cut close to the scalp 6 months after start of study participation (baseline - IUD insertion) to assess change from baseline to 6 months.

SECONDARY OUTCOMES:
Mean change in hair cortisol concentration - 12 months | Baseline & 12 months post-insertion
  A hair sample of approximately 10 (up to 20) hairs cut close to the scalp 12 months after start of study participation (baseline - IUD insertion) to assess change from baseline to 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Doty, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Doty N, Beckley E, Garg B, Maristany S, Erikson DW, Jensen JT. Changes in hair cortisol concentration in intrauterine device initiators: A prospective cohort study. Contraception. 2023 Dec;128:110142. doi: 10.1016/j.contraception.2023.110142. Epub 2023 Aug 24. PMID 37633589